CLINICAL TRIAL: NCT05640947
Title: Endoscopic Ultrasound-guided Large Diameter Lumen-apposing Metal Stent Gastro-gastrostomy for Bypass Reversal in Patients With Roux-en-y Gastric Bypass: a Proof of Concent Study
Brief Title: Endoscopic Ultrasound-guided Large Diameter Lumen-apposing Metal Stent Gastro-gastrostomy for Bypass Reversal in Patients With Roux-en-y Gastric Bypass
Acronym: LABOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2022-0015
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Hypoglycemia; Gastric Outlet Obstruction; Steatohepatitis; Parenteral Support; Gastric Bypass
MeSH Terms: conditions — Hypoglycemia; Gastric Outlet Obstruction; Fatty Liver

STUDY DESIGN:
Intervention Model Description: Placement of a 20mm lumen-apposing metal stent (Hot AxiosR, Boston Scientific) between the gastric pouch or the jejunum and the excluded stomach. The procedure will be performed by a physician with sufficient experience in the technique (more than 30 lumen-apposing metal stent placements of which more than 5 gastro-gastrostomies, the latter being the procedure that will be performed for the study). The proximal flange of the LAMS is preferably placed in the blind jejunal loop or, if this is not feasible, at least as far as possible from the gastro-oesophageal junction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- LAMS gastro-gastrostomy (Experimental)
  Interventions: Device: The Hot AXIOS™ Stent and Electrocautery-Enhanced Delivery System

INTERVENTIONS:
Device: The Hot AXIOS™ Stent and Electrocautery-Enhanced Delivery System — EUS-guided gastro-gastrostomy using the Hot Axios device: Using a therapeutic endoscopic ultrasound endoscope with a working channel of 3.7mm and under fluoroscopic control, the excluded stomach will be identified and punctured with a 19G needle. Contrast injection will confirm the good position of the needle in the excluded stomach. If needed, the excluded stomach will be filled with blue-stained aqua (5% indigocarmine) until a sufficient distension is obtained for placement of the lumen-apposing metal stent. A lumen-apposing metal stent with a diameter of 20mm will be used according to the manufacterers' instructions to create a gastrogastrostomy. Position will be checked with fluoroscopy.
  Other Names: LAMS

SUMMARY:
The primary objective of this open-label pilot study is to investigate whether an endoscopically placed lumen apposing metal stent is an effective alternative to surgery in patients that have a clear indication for reversal of their gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* Group 1) patients needing any kind of parenteral nutritional support (eg. hypo- albuminemia, hypovitaminoses, mineral deficiencies,...) that can not be corrected by dietary intervention/oral supplementation
* Group 2) patients with persistent invalidating symptomatic dumping syndrome despite optimal dietary intervention (typical complaints are headache, sweating, trembling, weakness and feeling hungry).
* Group 3) patients with a refractory marginal ulcers with stenosis of the gastrojejunostomy leading to feading difficulties.
* Group 4) patients with F3 or F4 liver fibrosis and a tendency to decompensation after bypass surgery, as demonstrated by an increase in serum bilirubin/INR and/or lowering of serum albumin.

Exclusion Criteria:

1. Uncorrectable coagulopathy
2. Presence of significant portal hypertension as demonstrated by 2.1) the presence of esophageal and/or gastric varices AND/OR 2.2) a hepatic venous pressure gradient (if measured) equal to or more than 10mm Hg AND/OR 2.3) the combination of

   1. a platelet count <150000/µl AND
   2. liver stiffness measured by elastometry equal to or more than 20 kPa (Baveno guidelines).
3. Pregnant women, breastfeeding women or women that can not assure adequate anticonception for the duration of the study (based on anamnesis).
4. Karnofsky index less than 60
5. Vulnerable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
clinical succes rate | 6 months
  1. for patients needing parenteral support: the number of parenteral supplements over a 6-month timeframe.
  2. for patients with symptomatic hypoglycemia: resolution of hypoglycemia- associated complaints + negative hypoglycemia-provocative testing (oral glucose tolerance test and/or mixed meal test) at 6 months post-intervention.
  3. for patients with gastric outlet obstruction: resolution of gastric outlet obstruction- associated symptoms at 6 months post-intervention.
  4. for patients with steatohepatitis and signs of liver failure: improvement of liver function (significant drop in bilirubin/INR; increase in serum albumin) at 6 months post-intervention.

SECONDARY OUTCOMES:
Technical success rate | 12 months
  Correct placement of the lumen-apposing metal stent in the desired position, scored yes/no
Duration of the procedure | 12 months
  time interval from scope introduction to successful deployment of the lumen-apposing metal stent.
Complication rate | 12 months
  These include procedure-related complications such as bleeding, perforation, stent migration, peritonitis, reflux disease … Complications will be divided into early (within 24h) and late (after 24h but within 30 days) complications.
  The severity of each complication will be scored as followed:
  1. mild: requiring admission or prolongation of planned admission <3 days;
  2. moderate: requiring prolongation of planned admission to 3-10 days;
  3. severe: requiring prolongation of planned admission to more than 10 days or requiring surgery;
  4. fatal: leading to death
Reintervention rate | 12 months
  endoscopic and/or surgical, reason should be clearly mentioned: due to loss of stent patency, stent migration, side-effects,…

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Hindryckx, Prof., Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - AZ Sint-Jan Brugge, Bruges
  - University Hospital, Ghent, Ghent

IPD SHARING:
Plan to Share IPD: No